# **Statistical Analysis Plan**

# SCR-004: Comprehensive *in vitro* Proarrhythmia Assay (CiPA) Clinical Phase 1 ECG Biomarker Validation Study

**Sponsor:** U.S. Food and Drug Administration

White Oak Building #64, Room 2072 10903 New Hampshire Avenue

Silver Spring, MD 20993

Sponsor Study Lead and Day

Medical Monitor:

David Strauss, MD, PhD

Director, Division of Applied Regulatory Science

U.S. Food and Drug Administration

Telephone: 301-796-6323

Email: david.strauss@fda.hhs.gov

FDA RIHSC Sponsor: David Strauss, MD, PhD

**Project Manager:** Jose Vicente, PhD

U.S. Food and Drug Administration

**Study Monitor:** Jill Brown

RIHSC Project Manager

U.S. Food and Drug Administration

Version of SAP: 5.1

Date of SAP: 25 March 2017

#### CONFIDENTIAL

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without the expressed written consent of the U.S. Food and Drug Administration.

## **Sponsor Signatures Page**

#### Prepared by

Jose Vicente Ruiz -S

Digitally signed by Jose Vicente Ruiz -S DN: c=US, o=U.S. Government, ou=HHS, ou=FDA, ou=People, 0.9.2342.19200300.100.1.1=2002160424, cn=Jose Vicente Ruiz -S Date: 2017.03.25 11:39:29 -04'00'

March 25, 2017

Date

Jose Vicente, PhD Visiting Scientist, Division of Cardiovascular and Renal Products U.S. Food and Drug Administration

#### Reviewed by

Robbert Zusterzeel - S cn-8 color 2017 03 25 11-45-52

Digitally signed by Robbert Zusterzeel -S DN: c=US, o=U.S. Government, ou=HHS, ou=FDA, ou=People, 0.9.2342.19200300.100.1.1=2001114905, Date: 2017.03.25 11:45:53 -04'00'

March 25, 2017 Date

Robbert Zusterzeel, MD, PhD Staff Fellow, Division of Applied Regulatory Science U.S. Food and Drug Administration

Approved by

Digitally signed by David Strauss -S DN: c=US, o=U.S. Government, ou=HHS, ou=FDA, ou=People, cn=David Strauss -S, 0.9.2342.19200300.100.1.1=2000507494 Date: 2017.03.25 14:01:10 -04'00'

March 25, 2017

Date

David Strauss, MD, PhD

Director, Division of Applied Regulatory

Science

U.S. Food and Drug Administration

# SCR-004: Comprehensive *in vitro* Proarrhythmia Assay (CiPA) Clinical Phase 1 ECG Biomarker Validation Study

## Contents

| Spo | nsor Sig | natures Page | 2 |
|---|---|---|---|
| Cor | itents | | 3 |
| 1 | Study C | Objectives | 6 |
| 1 | .1 Pri | mary Objective 1 (Part 1) | 6 |
| 1 | .2 Pri | mary Objective 2 (Part 2) | 6 |
| 2 | Sample | Size | 6 |
| 2 | .1 Re | sampling analysis methodology | 7 |
| 2 | .2 Par | rt 1 | 8 |
| 2 | .3 Par | rt 2 | 9 |
| 2 | .4 Re | placement Algorithm for Parts 1 and 2 | 10 |
| | 2.4.1 | Crossover part (Part 2): | 11 |
| | 2.4.2 | Parallel part (Part 1): | 12 |
| 3 | Analysi | is Populations | 15 |
| 4 | Genera | Statistical Considerations, Subject Disposition and Demographics and Baseline | • |
| Cha | racterist | ics | 15 |
| 5 | Electro | cardiogram Analyses | 16 |
| 5 | .1 An | alysis and removal of heart rate dependency for QT and J-T <sub>peak</sub> | 16 |
| 5 | .2 Pri | mary Analyses | 17 |
| | 5.2.1 | Parts 1 and 2 | 17 |
| | 5.2.2 | Part 1 | 18 |
| | 5.2.3 | Part 2 | 19 |
| 5 | .3 Ex | ploratory Analyses | 20 |
| | 5.3.1 | Exposure-response analysis of secondary ECG biomarkers | 20 |
| | 5.3.2 | $\Delta\Delta ECG$ measurements by time point | 20 |
| | 5.3.3 | Analyses using population-based heart rate corrected QT and J-Tpeak | 21 |
| | 5.3.4 | Use of placebo from parallel part in crossover part | 21 |
| 6 | Pharma | cokinetic Analyses | 22 |
| 7 | Safety A | Analyses | 22 |
| 8 | Missing | Data | 23 |

# Statistical Analysis Plan

# SCR-004: Comprehensive *in vitro* Proarrhythmia Assay (CiPA) Clinical Phase 1 ECG Biomarker Validation Study

| 9 Data Q | uality Assurance | 23 |
|---|---|---|
| 10 Refe | rences | 24 |
| A Randomi | zation schedule | 25 |
| A.1 Al | ostract | 25 |
| A.2 St | ndy design (pre-specified balanced design within period/cohort) | 26 |
| A.3 Tr | eatment codes and subjects IDs from 3 blocks by Part and Cohort | 26 |
| A.4 Ra | ndomization | 31 |
| A.4.1 | Seed random number generator | 31 |
| A.4.2 | Randomization schedule code | 31 |
| A.5 Fo | r clinical site unblinded pharmacist | 32 |
| A.5.1 | The random generator seed was: 123456 | 32 |
| A.5.2 | Randomized treatment codes | 32 |
| A.5.3 | Randomization schedule table | 33 |
| A.5.4 | Randomized summary table | 35 |
| A.6 Ap | pendix: technical information | 36 |
| B Step by s | tep example of replacement algorithm | 37 |
| B.1 Re | placement in crossover part | 37 |
| B.1.1 | Move RANDIDs from completers to the next period | 37 |
| B.1.2 | Replace dropouts | 38 |
| B.2 Re | placement in parallel part | 40 |
| B.2.1 | Step 1: (replace subject 1014 from placebo) | 41 |
| B.2.2 | Step 2: (replace subject 1002 from ranolazine) | 41 |
| B.2.3 | Step 3: (replace subject 1004 from verapamil) | 42 |
| B.2.4 | Step 4: (replace subject 1011 from chloroquine) | 42 |
| B.2.5 | Step 5: (replace subject 1007 from lopinavir+ritonavir) | 43 |
| B.2.6 | Step 6: (replace subject 1028 from placebo) | 43 |
| B.2.7 | Step 7: (replace subject 1018 from ranolazine) | 43 |
| B.2.8 | Step 8: (replace subject 1019 from verapamil) | 44 |
| B.2.9 | Step 9: (replace subject 1025 from chloroquine) | 44 |
| B.2.10 | Step 10: (replace subject 1024 from lopinavir+ritonavir) | 45 |

| Statistical A | Analysis Plan | SCR-004: Comprehensive <i>in vitro</i> Proarrhy (CiPA) Clinical Phase 1 ECG Biomarker Valid | |
|---|---|---|---|
| B.2.11 | Step 11: End (m | aximum number of 14 replacements reached) | 45 |

### 1 Study Objectives

The primary objectives of this study are:

- To confirm that exposure-response analysis of the electrocardiographic QTc and J-T<sub>peakC</sub> intervals in Phase 1 clinical pharmacology studies can be used to confirm that "balanced ion channel" drugs do not cause J-T<sub>peakC</sub> prolongation and "predominant hERG" drugs cause QTc prolongation.
- 2. To test the hypothesis that calcium channel block (diltiazem) can reduce the QTc prolongation from hERG block (dofetilide) by shortening J-T<sub>peakC</sub>.

## 1.1 Primary Objective 1 (Part 1)

Part 1 of the study will assess primary objective 1. Part 1 will include 4 oral drugs with well-characterized ion channel effects, QTc effects, and torsade de pointes (TdP) risk. Three (3) drugs will be "balanced ion channel" blockers (approximately equipotent hERG and late sodium and/or calcium block) with low TdP risk (ranolazine, verapamil and lopinavir + ritonavir) and 1 drug will be a "predominant hERG" blocker with TdP risk (chloroquine).

## 1.2 Primary Objective 2 (Part 2)

Part 2 of the study will assess primary objective 2. Part 2 will include 2 oral drugs (dofetilide and diltiazem) with well-characterized individual ion channel effects and TdP risk. Dofetilide is a "predominant hERG" blocker while diltiazem is a calcium channel blocker.

## 2 Sample Size

Approximately 60 healthy subjects are planned for enrollment, of which 50 will be assigned to Part 1 and 10 will be assigned to Part 2 at randomization. Up to 14 subjects may be qualified as replacements. Thus, a maximum of 74 subjects will be exposed to study drugs and procedures during the study.

The sample size (10 subjects per arm) was selected based on analysis by the sponsor of ECG biomarkers in Studies SCR-002<sup>1</sup> and SCR-003<sup>2</sup> and by resampling of data from previously conducted thorough QT (TQT) clinical studies, similar to the methodology of Ferber et al.<sup>3,4</sup> The data sources<sup>5,6</sup> used in this analysis are appropriate to determine the sample size because (i) the inclusion and exclusion criteria of this study are similar to inclusion and exclusion criteria in SCR-002, SCR-003 and typical TQT studies; (ii) this study will be conducted at the same clinical site than SCR-002 and SCR-003; (iii) the ECG analysis will be performed at FDA using the same methodology used in SCR-002 and SCR-003; and (iv) we observed consistent druginduced ECG signatures between SCR-002 and SCR-003 (Figure 1 and Figure 2).<sup>7</sup>



**Figure 1**. ECG signatures of predominant hERG block with dofetilide in both SCR-002 (Study 1, dark grey) and SCR-003 (Study 2, light grey) and with moxifloxacin in SCR-003 (yellow). Vicente et al. 2016.<sup>7</sup>



**Figure 2**. ECG signatures of multichannel block with ranolazine in SCR-002 (Study 1, blue) and dofetilide+lidocaine (green) and dofetilide+mexiletine (orange) vs. predominant hERG block with dofetilide alone (gray) in SCR-003 (Study 2). Vicente et al. 2016.<sup>7</sup>

## 2.1 Resampling analysis methodology

The overall methodology in this analysis is based on work by Ferber et al.,<sup>3,4</sup> where data from TQT studies is bootstrapped using sampling without replacement, likely due to the resampling size << number of subjects in the study, under different conditions: number of subjects on active drug and number on placebo. In the case of cross-over studies, subjects in either placebo or on active are treated as two different subjects, and the data is modeled using the following model (for QTc):

$$\Delta QTc_{i,j} = Treat_{i,j} + Time_{i,j} + \alpha_i Conc_{i,j} + \beta + \beta_i + \varepsilon_{i,j}$$

where subscripts i and j refer to subject ith measurement jth,  $\alpha$  is the slope,  $\beta$  is the intercept and there is a random effect on both the intercept and slope, and the random effects and the error term are assumed to be independent and identically distributed (i.i.d) normal. Of note, all time points are included in the analysis.

In our analysis, we bootstrapped the data from SCR-002 and SCR-003 using sampling with replacement because the number of subjects in these studies (22 subjects in each study) was similar to the sample size of the largest sample size of the simulated studies (from 6 to 24 subjects).

#### 2.2 Part 1

To estimate the sample size required to meet the endpoint of Part 1, we used data from a "predominant hERG" blocking drug (moxifloxacin from SCR-003), a "balanced ion channel" drug (ranolazine from SCR-002) and placebo (from both SCR-002 and SCR-003). We simulated 1000 parallel studies for each drug + placebo and scenario ranging from 3 subjects on placebo and 3 subjects on drug to 10 subjects on placebo and 14 subjects on drug (i.e. 160,000 studies). We bootstrapped the data using sampling with replacement because the number of subjects in these studies (22 subjects in each study) was similar to the sample size of the largest sample size of the simulated studies (up to 24 subjects). The results of resampling analysis suggest that 9 subjects on active study drug and 6 subjects on placebo will be sufficient to detect QTc prolongation for the "predominant hERG" drug and exclude J-T<sub>peakC</sub> prolongation for the "balanced ion channel" drugs (Figure 3). Figure 3 below shows simulation results using data from our previous studies and the following model using the lme4 package in R:

#### CHG~TPT+TRTA+CONC+(1+CONC|RANDID)

where CHG is change from baseline in the ECG biomarker (e.g.  $\Delta$ QTc), CONC is the drug concentration (set to 0 for placebo), TPT is time, TRT is the treatment (coded as 0 for placebo, 1 for active drug) and USUBJID is the subject identifier.

Due to the long half-life of some drugs that are included in this study and the desire to more closely mimic SAD/MAD studies, Part 1 of the current clinical study will use an entirely parallel study design with 10 subjects in each arm. Specifically, fifty (50) healthy subjects will be enrolled. Multiple doses of each drug will be given to 40 subjects on 3 consecutive days to achieve low and high exposures on Days 1 and 3, respectively, and 10 subjects will receive placebo.

It is anticipated that this study will be completed in 3 cohorts with approximately equal numbers of subjects per cohort. Cohorts 1 and 2 will have 15 subjects each (3 subjects per arm). Cohort 3 will have 20 subjects (4 subjects per arm). Up to 14 replacement subjects may be added to Cohort 3 if it is estimated that fewer than 8 subjects will complete the study in a study arm

following the replacement algorithm specified under "2.4 Replacement Algorithm for Parts 1 and 2".



**Figure 3**. Percentage of studies correctly classified as a function of the number of subjects on active drug with 6 subjects on placebo for (a) a hERG blocker (moxifloxacin) with QTc>=10ms; and (b) a "balanced ion channel" blocker (ranolazine) with J-T<sub>peakC</sub> < 10 ms.

#### 2.3 Part 2

To estimate the sample size required to meet the endpoint of Part 2, we used data from a "predominant hERG" blocking drug alone (dofetilide from SCR-003) and in combination with an inward current blocker (mexiletine from SCR-003). We simulated 1000 crossover studies for each scenario ranging from 3 to 10 subjects completing the study (i.e. 8,000 studies = 8 different sample sizes x 1000 simulations). We bootstrapped the data using sampling with replacement because the number of subjects in study SCR-003 (10 subjects in the each treatment sequence) was equal to the sample size of the largest sample size of the simulated studies (up to 10 subjects). The results of resampling analysis demonstrated that inward current block (mexiletine) effects on the QTc and J-T<sub>peakC</sub> slopes could be detected approximately 99% and 99% of the time, respectively, using a crossover design with 8 subjects (i.e., the inward current blocker (mexiletine) significantly reduced prolongation from the hERG blocker (dofetilide)). Figure 4 below shows simulation results using dofetilide and mexiletine data from our previous study SCR-003 and the following model using the lme4 package in R:

CHG~DOF+MEXI+DOF\*MEXI+(1+DOF|USUBJID)+(1+MEXI|USUBJID)

where CHG is change from baseline in the ECG biomarker (e.g.  $\Delta QTc$ ), DOF is the dofetilide concentration, MEXI is mexiletine concentration and USUBJID is the subject identifier.



**Figure 4:** Percentage of studies where late sodium blocker (mexiletine) significantly (p<0.05) reduced prolongation from the hERG blocker (dofetilide) for QTc (left panel) and for QTc first and then J-T<sub>peakC</sub> (right panel). Each sample size included 1,000 simulated studies using data from SCR-003 Vicente et al. 2016.<sup>7</sup>

Ten (10) healthy subjects will be enrolled for this part. Multiple doses of each drug (dofetilide and diltiazem) will be given either separately or together on 3 consecutive days in the first period and again on 3 consecutive days in the second period, depending on the randomization, to achieve low and high exposures on Days 1 and 3, respectively. There will be no placebo arm.

It is anticipated that Part 2 of this study will be completed in 1 cohort with 10 subjects with a crossover design. Similar to Part 1, subjects may be replaced in a later cohort if it is estimated that fewer than 8 subjects will complete Part 2. A maximum of 14 replacement subjects may be enrolled in the study.

## 2.4 Replacement Algorithm for Parts 1 and 2

Randomization identifiers for the potential replacements (REPLCMNTID) will be provided in the randomization schedule (see example in appendix A). The replacement algorithm to guide the unblinded Spaulding pharmacist is described below. A step by step example is provided in appendix B.

#### 2.4.1 Crossover part (Part 2):

After Period 1 and before check-in of Period 2:

- 1. After period 1 assess number of dropouts in the crossover part (Part 2)
- 2. Allocate 1 replacement for each dropout up to 4 replacements to start on Period 2 together with those already participating.
  - a. If there are more than 4 dropouts, replacements will be done one subject per sequence at a time ordering dropouts by RANDID within sequence and starting with the lowest RANDID (example in appendix A).

Flow-chart of management of replacements for the crossover part. Assessment will be done after Period 1 and before check-in of Period 2



Nxo: Number of dropouts in the crossover part in Period 1 (i.e. before Period 2 check-in).

#### 2.4.2 Parallel part (Part 1):

Parallel part (Part 1) will be assessed after its second cohort (Cohort 3) finishes and before the check-in of its last cohort (Cohort 4):

- 1. After the second cohort of the parallel part (Cohort 3) finishes assess number of dropouts in the parallel part (Part 1)
- 2. Replace each dropout up to the maximum number of 14 for the whole study (Parts 1 and 2 together). If the maximum will be reached, prioritize which treatment arms will receive replacements to bring the total number of completers in a treatment arm closer to 10 in the following order: 1) placebo, 2) ranolazine, 3) verapamil, 4) chloroquine, 5) lopinavir/ritonavir. For example, first bring all arms up to having at least 9 subjects per arm, and then if there are 2 remaining potential replacements, allocate them to placebo and ranolazine (see flow chart for parallel part in following pages and example in appendix B).

Flow-chart of management of replacements for the parallel part. Assessment will be done after the second cohort (Cohort 3) finishes and before the check-in of the last cohort (Cohort 4) of the parallel part





Page 14 of 45

Table of acronyms in the flow chart:

| Acronym | Description |
|---|---|
| Nrpl | Number of replacement that are available (i.e. how many of the 14 potential |
| | replacements have not been allocated yet) |
| C1Cpbo | Number of subjects that completed Cohort 1 of placebo arm |
| C3Cpbo | Number of subjects that completed Cohort 3 of placebo arm |
| Rpbo | Number of replacements allocated to the ranolazine arm |
| C1Cran | Number of subjects that completed Cohort 1 of ranolazine arm |
| C3Cran | Number of subjects that completed Cohort 3 of ranolazine arm |
| Rran | Number of replacements allocated to the ranolazine arm |
| C1Cver | Number of subjects that completed Cohort 1 of verapamil arm |
| C3Cver | Number of subjects that completed Cohort 3 of verapamil arm |
| Rver | Number of replacements allocated to the verapamil arm |
| C1Cchl | Number of subjects that completed Cohort 1 of chloroquine arm |
| C3Cchl | Number of subjects that completed Cohort 3 of chloroquine arm |
| Rchl | Number of replacements allocated to the chloroquine arm |
| C1Clvrv | Number of subjects that completed Cohort 1 of lopinavir+ritonavir arm |
| PC3Clvrv | Number of subjects that completed Cohort 3 of lopinavir+ritonavir arm |
| Rlvrv | Number of replacements allocated to the lopinavir+ritonavir arm |

## 3 Analysis Populations

The exposure-response population will include all subjects who receive at least 1 dose of any of the study drugs and have digital ECG (QTc and J-T<sub>peakC</sub>) data for the treatment period collected before dosing and at 1 or more time points after dosing as well as plasma concentration data (except for the placebo arm) from the same time points after dosing. Subjects in this population will be used for the exposure-response analysis.

The PK population will include all subjects who receive study drug and have at least 1 estimable PK parameter after dosing.

The safety population will include all subjects who receive at least 1 dose of any of the study drugs.

## 4 General Statistical Considerations, Subject Disposition and Demographics and Baseline Characteristics

All data will be presented in data listings. Data from subjects excluded from an analysis population will be presented in the data listings but not included in the calculation of summary statistics. The number of subjects who enroll in the study and the number and percentage of

subjects who complete each assessment will be presented. The frequency and percentage of subjects who withdraw or discontinue from the study and the reason for withdrawal or discontinuation will be summarized. Continuous demographic and baseline characteristic variables (age, height, weight, body mass index) will be summarized overall and by treatment using descriptive statistics (number of subjects, mean, standard deviation [SD], median, and minimum and maximum). The number and percentage of subjects in each class of categorical demographic and baseline characteristic variables will also be summarized.

## 5 Electrocardiogram Analyses

### 5.1 Analysis and removal of heart rate dependency for QT and J-T<sub>peak</sub>

For the primary analysis, the QT interval will be corrected for heart rate using Fridericia's formula (QTc=QT/RR<sup>1/3</sup>). The J-T<sub>peak</sub> interval will be corrected for heart rate using the Johannesen et al  $(2014)^8$  formula (J-T<sub>peakC</sub> = J-T<sub>peakC</sub>/RR<sup>0.58</sup>).

If any drug causes an absolute placebo corrected change from baseline in heart rate ( $\Delta\Delta$ HR) greater than 10 beats per minute (i.e. mean effect >10bpm change in either direction) at any time point, then we will assess goodness of HR correction (visual assessment on plots like the example ones in Figure 5):

- 1. QT vs RR and QTcF vs RR
- 2.  $J-T_{peak}$  vs RR and  $JT_{peak}$ C vs RR



**Figure 5**: Example of plots for assessing goodness of HR correction. QT and RR data from placebo arm and baseline time points from SCR-003.

If there are HR effects >10 bpm and the relationship does not look appropriate (per visual assessment) then we will perform an analysis using population-based HR correction (described below).

## 5.2 Primary Analyses

Analysis flow chart (for each endpoint):



#### 5.2.1 Parts 1 and 2

Investigation of hysteresis: Prior to model selection for the exposure-response analysis, the presence of hysteresis will be assessed for QTc and J- $T_{peakC}$ . To detect hysteresis, individual change-from-baseline in J- $T_{peakC}$  ( $\Delta J$ - $T_{peakC}$ ) will be computed. For each day, the time of the largest mean  $\Delta J$ - $T_{peakC}$  ( $U_{max}$ ) will be determined. If the largest mean  $\Delta J$ - $T_{peakC}$  exceeds 5 msec at  $\geq$ 3 time points, the time difference between  $U_{max}$  and the  $T_{max}$  of the drug level exceeds 1 hour, and the 1-sided, 1-sample Wilcoxon test for the difference between  $\Delta J$ - $T_{peakC}$  at  $T_{max}$  and at  $U_{max}$  is formally significant at the 1% level, it will be concluded that hysteresis existed. In such a case, a PK model with an additional effect compartment will replace the model described below. The same steps will be followed for QTc as part of the primary endpoint.

<u>Model selection</u>: To assess the appropriateness of a linear model, normal QQ-plots for the residuals and plots of weighted residuals versus concentration and versus fitted values will be produced. A model with a quadratic term in concentration will be fitted and the quadratic term will be tested on the 2-sided 5% alpha level. If there is a significant quadratic term, nonlinear models, such as a log-linear model and an  $E_{max}$  model, will be investigated and the primary

model will be selected based on the Akaike Information Criterion (AIC) and plausibility arguments.

Exposure-response analysis: In the absence of hysteresis and unless the pre-specified test procedure for linearity indicates otherwise, the primary analysis will be based on a linear mixed-effects model implemented in SAS® or R software, with  $\Delta J$ -T<sub>peakC</sub> as the dependent variable, drug plasma concentration as continuous covariate, treatment and time point as categorical factors, and subject-specific random effects for the intercept and slope, depending on whether Part 1 or Part 2 of the study is being considered (details for each part below). All postdose data will be used. The degrees of freedom for the model estimates will be determined by the Kenward-Rogers method. From the model, the slope (i.e., the regression parameter for the concentration) and the treatment effect will be estimated together with 2-sided 90% CIs.

The predicted mean placebo-adjusted change-from-baseline J- $T_{peakC}$  ( $\Delta\Delta J$ - $T_{peakC}$ ) at the observed geometric mean  $C_{max}$  (i.e., the product with the slope estimate + treatment effect [ $\Delta J$ - $T_{peakCactive}$  –  $\Delta J$ - $T_{peakCplacebo}$ ]) and the 2-sided 90% CI of the estimate will be calculated. The same steps will be followed for QTc as part of the primary endpoint.

#### 5.2.2 Part 1

The primary variable for the exposure-response analysis will be the change-from-baseline in QTc ( $\Delta QTc$ ) for the "predominant hERG" drug and change-from-baseline in J-T<sub>peakC</sub> ( $\Delta J$ -T<sub>peakC</sub>) for the "balanced ion channel" drugs, where the mean of the 3 predose ECG readings on Day 1 will be used as the Baseline. The concentration of the drug will be used as a covariate. Exposure-response analysis will be done following most recent best practices in concentration-QTc modeling.

#### Criteria for primary QTc and J-T<sub>peakC</sub> assessment:

Criteria for the 3 "balanced ion channel" drugs (ranolazine, verapamil, lopinavir + ritonavir) will be based on the predicted J-T<sub>peakC</sub> effect on the third day of dosing. To demonstrate a lack of placebo-adjusted change-from-baseline J-T<sub>peakC</sub> ( $\Delta\Delta$ J-T<sub>peakC</sub>) prolongation for each of the 3 drugs:

- The upper bound of the 2-sided 90% CI of the predicted mean  $\Delta\Delta J$ -T<sub>peakC</sub> must be <10 msec at the observed geometric mean C<sub>max</sub> on Day 3.
  - o  $H_0$ :  $\Delta \Delta J$ - $T_{peakC} \ge 10 \text{ ms}$
  - $\circ \quad H_{\text{A}}\!\!:\Delta\Delta J\text{-}T_{\text{peakC}}\!<10\;ms$

Criteria for the "predominant hERG" drug (chloroquine) will be based on the predicted QTc effect on the first day of dosing. To demonstrate the presence of placebo-adjusted change-from-baseline QTc ( $\Delta\Delta$ QTc) prolongation for chloroquine:

# SCR-004: Comprehensive *in vitro* Proarrhythmia Assay (CiPA) Clinical Phase 1 ECG Biomarker Validation Study

- The upper bound of the 2-sided 90% CI of the predicted mean ΔΔQTc must be ≥10 msec at the observed geometric mean C<sub>max</sub> on Day 1.
  - $\begin{array}{ll} \circ & H_0\text{: } \Delta\Delta QTc \leq 10 \text{ ms} \\ \circ & H_\text{A}\text{: } \Delta\Delta QTc \geq 10 \text{ ms} \\ \end{array}$

We will use the following linear mixed effects model (QTc as example):

$$\Delta QTc \sim time + treatment + concentration + (1+concentration|subjid)$$

where concentration is set to 0 for placebo, treatment is 1 for drug and 0 for placebo, and time is a categorical variable coded as time after first dose (e.g. '1 hr', 1.5 hr', '2 hr', '4 hr', ... '72 hr'). Note that the prediction from the model above is  $\Delta\Delta QTc$  because placebo treatment is coded as 0

In addition to the tests specified above (e.g.  $\Delta\Delta QTc \ge 10$  ms at Cmax of Day 1), it will be assessed:

- 1. whether exploratory plots suggest model misspecification
  - a. Exploratory plot will show the model fit (mean and 95%CIs) plot on top of the observed  $\Delta\Delta QTc$  ( $\Delta QTc_{drug}$  mean  $\Delta QTc_{placebo}$  by time) and the corresponding deciles of the observed data
  - b. QQ-plots of the model residuals
  - c. Plot of the standardized residuals by time, treatment and concentration (continuous for continuous variables, otherwise boxplot)

If there is an effect (e.g.  $abs(\Delta\Delta QTc) \ge 10$  ms) and the fit is acceptable then we accept the linear model. If not (i.e. either or both criteria are not met) then further models will be assessed. The same assessment will be performed for J-Tpeakc in a similar fashion.

#### 5.2.3 Part 2

The primary variable for the exposure-response analysis will be the change-from-baseline in QTc ( $\Delta$ QTc) for the pooled dofetilide alone, diltiazem alone, and dofetilide + diltiazem, where the mean of the 3 predose ECG readings on Day 1 will be used as the Baseline. The concentration of dofetilide and diltiazem will be used as covariates.

## Criteria for primary QTc and J-T<sub>peakC</sub> assessment:

To demonstrate that calcium channel block (diltiazem) reduces QTc prolongation from hERG block (dofetilide) by shortening J-T<sub>peakC</sub>:

• It will be assessed whether the projected QTc effect of dofetilide alone is significantly greater (i.e., p<0.05) than the projected QTc effect of the combination of dofetilide +

# SCR-004: Comprehensive *in vitro* Proarrhythmia Assay (CiPA) Clinical Phase 1 ECG Biomarker Validation Study

diltiazem. This will be assessed at the dofetilide peak plasma level on Day 3 (computed from the combination of dofetilide + diltiazem) on the pooled dofetilide alone, diltiazem alone, and dofetilide + diltiazem data using a linear mixed effects model:

- ΔQTc ~ DOF+DILT+DOF\*DILT+(1+DOF| USUBJID)+(1+DILT| USUBJID)
   where DOF is concentration of dofetilide, and DILT is concentration of diltiazem.
  - $H_0$ :  $\triangle QTc$  (Dof Cmax, Dilt=0)  $\leq \triangle QTc$  (Dof Cmax, Dilt Cmax)
  - $H_A$ :  $\triangle QTc$  (Dof Cmax, Dilt=0)  $> \triangle QTc$  (Dof Cmax, Dilt Cmax)
- If the previous test is statistically significant for QTc, the same test will be performed for J-Tpeakc.
  - $\circ \quad \Delta JTpeakc \sim DOF + DILT + DOF * DILT + (1 + DOF \mid USUBJID) + (1 + DILT \mid USUBJID)$ 
    - H<sub>0</sub>: ΔJTpeakc (Dof Cmax, Dilt=0) ≤ ΔJTpeakc (Dof Cmax, Dilt Cmax)
    - H<sub>A</sub>: ΔJTpeakc (Dof Cmax, Dilt=0) > ΔJTpeakc (Dof Cmax, Dilt Cmax)

In addition to the tests specified above, it will be assessed:

- 1. whether exploratory plots suggest model misspecification
  - a. Exploratory plot will show the model fit (mean and 95%CIs) plot on top of the observed  $\Delta QTc$  and the corresponding deciles of the observed data.
  - b. QQ-plots of the model residuals
  - c. Plot of the standardized residuals by time, treatment and concentration (continuous for continuous variables, otherwise boxplot)

If there is a  $\triangle QTc$  effect and the fit is acceptable then we accept the linear model. If not (i.e. either or both criteria are not met) then further models will be assessed. The same assessment will be performed for J-Tpeakc in a similar fashion.

## 5.3 Exploratory Analyses

## 5.3.1 Exposure-response analysis of secondary ECG biomarkers

Exposure-response analysis of secondary ECG biomarkers: For Part 1, exposure-response analysis similar to that described for QTc and J-T<sub>peakC</sub> will be applied to PR, QRS, QTc, J-T<sub>peakC</sub>, and T<sub>peak</sub>-T<sub>end</sub> for Day 1 and Day 3. This will also include analysis of change from baseline for dofetilide alone, diltiazem alone, and dofetilide + diltiazem combination from Part 2 of the study.

#### **5.3.2** ΔΔECG measurements by time point

For each time point, an analysis of variance model will be fitted with  $\Delta J$ - $T_{peakC}$  as the dependent variable, treatment (active or placebo) as factor, and baseline J- $T_{peakC}$  as a covariate. From this

model, the difference ( $\Delta J$ -T<sub>peakCactive</sub> –  $\Delta J$ -T<sub>peakCplacebo</sub>) will be estimated with a 2-sided 90% CI. Separate models will be fitted for each treatment, all of them using the same placebo data. The same steps will be followed for QTc. Change from Baseline in heart rate, PR, QRS, and T<sub>peak</sub>-T<sub>end</sub> will be calculated using descriptive summary statistics.

#### 5.3.3 Analyses using population-based heart rate corrected QT and J-Tpeak

If any drug causes an absolute placebo-corrected change from baseline in heart rate greater than 10 beats per minute, we will perform exposure-response and  $\Delta\Delta ECG$  measurements by time point using population-based heart rate correction factors for OT and J-Tpeak. We will use continuous/Holter 12-lead ECGs recorded at check-in from early afternoon until the subjects go to sleep. During this period, subjects will perform a sequence of postural maneuvers (e.g., 10 minutes supine, 10 minutes sitting, 10 minutes standing, 10 minutes sitting, 10 minutes supine) to characterize ECG biomarkers and heart rate relationship (i.e. QT/RR and J-T<sub>peak</sub>/RR relationships). From each Holter and postural maneuver window, triplicate 10-second 12-lead ECGs will be extracted at different heart rates. Additional details will be available in the ECG analysis plan. The dependency of the different electrocardiographic intervals on heart rate will be evaluated using the extracted ECGs from the Holters. We will compute a population-based correction factor using an exponential model. The model will include random effects for the intercept  $(\log(\alpha))$  and  $\beta$  (i.e., allowing each individual to have his or her own slope). We will consider that there is heart rate dependency for an ECG biomarker if the ECG biomarker and heart rate relationship is significant and there is at least 10% of change in the ECG biomarker within the heart rate range as described in Johannesen et al 2014.8 For heart rate dependent ECG biomarkers, the individual correction factors will be applied using the exponential model. Using QT as an example:  $QTcI = QT/RR^{\beta i}$ , where  $\beta i$  is the slope of the relationship of the i-th subject.

#### 5.3.4 Use of placebo from parallel part in crossover part

The 10-subject placebo group from the parallel part of the study can potentially be used interchangeably with the crossover part. This analysis will test that calcium channel block (diltiazem) reduces QTc prolongation from hERG block (dofetilide) by shortening J-T<sub>peakC</sub>. The placebo corrected changes from baseline ( $\Delta\Delta$ ) will be computed subtracting the time-matched average placebo changes from baseline ( $\Delta$ ) of the subjects participating in Part 1 of the study from the individual changes from baseline of subjects participating in Part 2.

- It will be assessed whether the projected QTc effect of dofetilide alone is significantly greater (i.e., p<0.05) than the projected QTc effect of the combination of dofetilide + diltiazem. This will be assessed at the dofetilide peak plasma level on Day 3 (computed from the combination of dofetilide + diltiazem) on the pooled dofetilide alone, diltiazem alone, and dofetilide + diltiazem data using a linear mixed effects model using the placebo-corrected change from baseline as dependent variable:
  - $\bigcirc \quad \Delta \Delta QTc \sim DOF + DILT + DOF *DILT + (1 + DOF \mid USUBJID) + (1 + DILT \mid USUBJID)$

where DOF is concentration of dofetilide, and DILT is concentration of diltiazem.

- $H_0$ :  $\Delta\Delta QTc$  (Dof Cmax, Dilt=0)  $\leq \Delta\Delta QTc$  (Dof Cmax, Dilt Cmax)
- $H_A$ :  $\Delta\Delta QTc$  (Dof Cmax, Dilt=0) >  $\Delta\Delta QTc$  (Dof Cmax, Dilt Cmax)
- If the previous test is statistically significant for QTc, the same test will be performed for J-Tpeakc.
  - $\circ \quad \Delta \Delta JTpeakc \sim DOF + DILT + DOF *DILT + (1 + DOF \mid USUBJID) + (1 + DILT \mid USUBJID)$ 
    - $H_0$ :  $\Delta\Delta JT$  peaks (Dof Cmax, Dilt=0)  $\leq \Delta\Delta JT$  peaks (Dof Cmax, Dilt Cmax)
    - H<sub>A</sub>: ΔΔJTpeakc (Dof Cmax, Dilt=0) > ΔΔJTpeakc (Dof Cmax, Dilt Cmax)

## 6 Pharmacokinetic Analyses

PK parameters C<sub>max</sub>, T<sub>max</sub>, and AUC will be summarized using descriptive statistics (number of subjects, mean, standard deviation [SD], coefficient of variation [CV], median, minimum, and maximum) for Day 1 and Day 3 for each active drug and period (i.e., Days 1 and 3 of Part 1 and Days 1, 3, 8 and 10 of Part 2). The PK parameters will be analyzed using non-compartmental methods based on actual sampling times. Mean and individual concentration-time profiles will be presented in graphs.

## 7 Safety Analyses

All AEs will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of treatment-emergent adverse events (TEAEs), organized by system organ class and frequency, will be summarized by seriousness, severity, relationship to treatment, and by treatment at onset of the TEAE. A detailed listing of serious AEs and TEAEs leading to withdrawal will also be provided.

Clinical laboratory results (hematology, serum chemistry, and urinalysis) will be summarized using descriptive statistics (number of subjects, mean, SD, minimum, median, and maximum). Clinical laboratory results will be classified as normal or abnormal, according to the reference ranges of the individual parameter. The number and percentage of subjects with abnormal laboratory results will be provided. No statistical testing will be performed on clinical laboratory data.

Vital sign measurements (blood pressure, heart rate, respiratory rate, and oral body temperature), safety 12-lead ECG results, and changes from Baseline for these parameters will be summarized by treatment and time point using descriptive statistics (number of subjects, mean, SD, minimum, median, and maximum). Physical examination findings will be presented in a data listing, and abnormal physical examination findings will be recorded as AEs.

All concomitant medication usage and medications that changed in daily dose, frequency, or both since the subject provided informed consent will be summarized for each subject.

### 8 Missing Data

Missing data will not be imputed. Data that are excluded from the descriptive or inferential analyses will be included in the subject data listings. This will include data from subjects not in the particular analysis population, measurements from unscheduled visits, or extra measurements that may arise from 2 or more analyses of a plasma sample at the same time point.

## 9 Data Quality Assurance

Completed eCRFs are required for each subject randomly assigned to study drug. Electronic data entry will be accomplished through the ClinSpark remote electronic data capture (EDC) system, which allows for on-site data entry and data management. This system provides immediate, direct data transfer to the database, as well as immediate detection of discrepancies, enabling site coordinators to resolve and manage discrepancies in a timely manner. Each person involved with the study will have an individual identification code and password that allows for record traceability. Thus, the system, and subsequently any investigative reviews, can identify coordinators, investigators, and individuals who have entered or modified records.

Furthermore, the investigator retains full responsibility for the accuracy and authenticity of all data entered into the electronic data capture system. The completed dataset and their associated files are the sole property of the sponsor and should not be made available in any form to third parties, except for appropriate governmental health or regulatory authorities, without written permission of the sponsor.

#### 10 References

- 1. Johannesen L, Vicente J, et al. Differentiating drug-induced multichannel block on the electrocardiogram: randomized study of dofetilide, quinidine, ranolazine, and verapamil. Clin Pharmacol Ther. 2014 Nov;96(5):549-58.
- 2. Johannesen L, Vicente J, et al. Late sodium current block for drug-induced long QT syndrome: Results from a prospective clinical trial. Clin Pharmacol Ther. 2016 Feb;99(2):214-23.
- 3. Ferber G, Zhou M, Darpo B. Detection of QTc effects in small studies--implications for replacing the thorough QT study. Ann Noninvasive Electrocardiol. 2015;20(4):368-77.
- 4. Ferber G, Lorch U, Taubel J. The Power of Phase I Studies to Detect Clinical Relevant QTc Prolongation: A Resampling Simulation Study. Biomed Res Int. 2015;2015:293564.
- 5. Vicente J, Johannesen L, Strauss DG. ECG Effects of Ranolazine, Dofetilide, Verapamil, and Quinidine in Healthy Subjects. doi:10.13026/C2HP45. url: https://physionet.org/physiobank/database/ecgrdvq/.
- 6. Vicente J, Johannesen L, Strauss DG. ECG effects of Dofetilide, Moxifloxacin, Dofetilide+Mexiletine, Dofetilide+Lidocaine and Moxifloxacin+Diltiazem in Healthy Subjects. doi:10.13026/C2D016. url: <a href="https://physionet.org/physiobank/database/ecgdmmld/">https://physionet.org/physiobank/database/ecgdmmld/</a>.
- 7. Vicente, J., L. Johannesen, M. Hosseini, J. W. Mason, P. T. Sager, E. Pueyo and D. G. Strauss (2016). "Electrocardiographic Biomarkers for Detection of Drug-Induced Late Sodium Current Block." PLOS ONE 11(12): e0163619.
- 8. Johannesen, L., J. Vicente, R. A. Gray, L. Galeotti, Z. Loring, C. E. Garnett, J. Florian, M. Ugander, N. Stockbridge and D. G. Strauss (2014). "Improving the assessment of heart toxicity for all new drugs through translational regulatory science." Clin Pharmacol Ther 95(5): 501-508.

#### A Randomization schedule

This code does not necessarily reflect any position of the Government or the Food and Drug Administration.

#### A.1 Abstract

This script generates the randomization schedule for the CiPA ECG clinical study (SCR-004).

After screening, 60 subjects will be randomized to participate in one of the 7 treatment sequences of the study. Example of treatment codes from the study protocol:

- Treatment sequences of Part 1 (parallel part)
  - A: Ranolazine (10 subjects)
  - B: Verapamil (10 subjects)
  - C: Lopinavir+Ritonavir (10 subjects)
  - D: Chloroquine (10 subjects)
  - E: Placebo (10 subjects)
- Treatment sequences of Part 2 (crossover part)
  - F,G: Dofetilide, Diltiazem+Dofetilide (5 subjects)
  - G,F: Diltaizem+Dofetilide, Dofetilide (5 subjects)

This script performs randomization in permuted blocks to achieve balance across treatment groups. The blocks are defined as follows:

- Block 1: First 15 subjects of parallel part (Cohort 1, Period 1) and 10 subjects of crossover part (Cohort 2, Periods 1 and 2)
  - Treatment sequences:
    - Parallel part: A, B, C, D, E
    - Crossover part: F-G, G-F
- Block 2: Second 15 subjects of parallel part (Cohort 3, Period 2)
  - Treatment sequences:
    - Parallel part: A, B, C, D, E
- Block 3: Remaining 20 subjects of parallel part (Cohort 4, Period 3)
  - Treatment sequences:
    - Parallel part: A, B, C, D, E

IDs for the potential replacements (REPLCMNTID) are computed from the randomization IDs (RANDID) as follows.

- In the parallel part (Part 1) REPLCMNTID = RANDID+2000
- In the crossover part (Part 2) there are 2 replacements (one per treatment sequence) for each drop out (up to 4 replacement total). Thus, each subject has two potential replacements IDs:

- For the replacement with same sequence than the dropout REPLCMNTID = 10\*(RANDID+2000) + 1 (e.g. 40011 for subject 2001)
- For the replacement with the alternative sequence than the dropout REPLCMNTID
   = 10\*(RANDID+2000) + 2 (e.g. 40012 for subject 2001)

#### A.2 Study design (pre-specified balanced design within period/cohort)

### A.3 Treatment codes and subjects IDs from 3 blocks by Part and Cohort

```
##
# List of randomization IDs
##
randids \leftarrow c(seq(1001, 1050, 1), seq(2001, 2010, 1))
##
# Randomization of treatment codes
treatmentcodespart1 <- c('A', 'B', 'C', 'D', 'E')
treatmentnamespart1 <- c('Ranolazine', 'Verapamil', 'Lopinavir+Ritonavir', 'Chlo</pre>
roquine','Placebo')
treatmentcodespart2 <- c('F','G')</pre>
treatmentnamespart2 <- c('Dofetilide', 'Diltiazem+Dofetilide')</pre>
##
# Treatment codes data.frame
##
treatments <- data.frame(CODE=c(treatmentcodespart1,treatmentcodespart2),TREA
TMENT=c (treatmentnamespart1, treatmentnamespart2), PART=c(1,1,1,1,1,2,2))
##
# Treatment sequences
part1seqs <- c('A', 'B', 'C', 'D', 'E')</pre>
part2seqs <- c('F-G','G-F')</pre>
##
# Block1
block1 \leftarrow data.frame(SEQ=c(part1seqs,part2seqs),NSUBJ=c(3,3,3,3,3,5,5),PART=
c(1,1,1,1,1,2,2), COHORT=c(1,1,1,1,1,2,2))
block1 <- block1 %>% group_by(PART) %>% mutate(CUMSUBJ=cumsum(NSUBJ)) %>% ung
roup()
block1 <- block1 %>% mutate(Group number=group indices(block1,.dots=c(SEQ)))
%>% group by(Group number) %>% mutate(RANDIDs=paste0(PART*1000+seq(CUMSUBJ-NS
UBJ+1,CUMSUBJ,1),collapse=', ')) %>% ungroup() %>% data.frame() %>% mutate(SE
Q=as.character(SEQ))
```

```
##
# Block2
block2 <- data.frame(SEQ=part1seqs,NSUBJ=3,PART=1,COHORT=3)</pre>
block2 <- block2 %>% group_by(PART) %>% mutate(CUMSUBJ=cumsum(NSUBJ)) %>% unq
roup()
block2 <- block2 %>% mutate(Group_number=group_indices(block2,.dots=c(SEQ)))
%>% group by(Group number) %>% mutate(RANDIDs=paste0(15+PART*1000+seq(CUMSUB
J-NSUBJ+1, CUMSUBJ, 1), collapse=', ')) %>% ungroup() %>% data.frame() %>% mutat
e(SEQ=as.character(SEQ))
##
# Block3
block3 <- data.frame(SEQ=part1seqs, NSUBJ=4, PART=1, COHORT=4)</pre>
block3 <- block3 %>% group_by(PART) %>% mutate(CUMSUBJ=cumsum(NSUBJ)) %>% ung
block3 <- block3 %>% mutate(Group number=group indices(block3,.dots=c(SEQ)))
%>% group by(Group number) %>% mutate(RANDIDs=paste0(30+PART*1000+seq(CUMSUB
J-NSUBJ+1,CUMSUBJ,1),collapse=', ')) %>% ungroup() %>% data.frame() %>% mutat
e(SEQ=as.character(SEQ))
##
# Schedule
schedule <- bind rows(block1, block2, block3) %>% select(-c(Group number, CUMS
UBJ,NSUBJ))
# Next statements were used during development to validate wide/long c
onversion operation
#schedule.summary <- schedule %>% spread(COHORT, RANDIDs)
#schedule.summary[is.na(schedule.summary)] <- ''</pre>
#pander(schedule.summary,split.table=Inf)
# Save schedule in long format to facitilate shuffle operations in the
randomization process below
schedulelong <- schedule %>% group_by(COHORT,SEQ) %>% mutate(ID1=strsplit(RAN
DIDs, ', ')[[1]][1], ID2=strsplit(RANDIDs, ', ')[[1]][2], ID3=strsplit(RANDIDs, ', ')
[[1]][3], ID4=strsplit(RANDIDs, ', ')[[1]][4], ID5=strsplit(RANDIDs, ', ')[[1]][5]
) %>% ungroup() %>% select(-RANDIDs) %>% gather(ID,RANDID,c(ID1,ID2,ID3,ID4,I
D5)) %>% filter(!is.na(RANDID)) %>% select(-ID) %>% distinct() %>% mutate(RA
NDID=as.numeric(RANDID)) %>% select(RANDID,PART,COHORT,SEQ) %>% arrange(RANDI
D)
# Schedule printed in section below
# pander(schedulelong,split.table=Inf)
```

```
#Format in summary table
schedulelong.summary <- schedulelong %>% group_by(COHORT,SEQ) %>% mutate(RAND
IDs=paste0(RANDID,collapse=', ')) %>% select(-RANDID) %>% ungroup() %>% disti
nct() %>% spread(COHORT,RANDIDs)
schedulelong.summary[is.na(schedulelong.summary)] <- ''

# Add potential replacements IDS to the long format
addpotentialreplacementids<-function(schdf){
   return (schdf %>% mutate(REPLCMNTID=RANDID+2000))
}
schedulelongwithrplids <- addpotentialreplacementids(schedulelong)
# Print table
# pander(schedulelong.summary,split.table=Inf)</pre>
```

#### A.3.1.1 Treatment codes

pander(treatments, split.table=Inf)

| CODE | TREATMENT | PART |
|------|----------------------|------|
| Α | Ranolazine | 1 |
| В | Verapamil | 1 |
| С | Lopinavir+Ritonavir | 1 |
| D | Chloroquine | 1 |
| E | Placebo | 1 |
| F | Dofetilide | 2 |
| G | Diltiazem+Dofetilide | 2 |

#### A.3.1.2 Treatment schedule

pander(schedulelongwithrplids ,split.table=Inf)

| RANDID | PART | COHORT | SEQ | REPLCMNTID |
|--------|------|--------|-----|------------|
| 1001 | 1 | 1 | Α | 3001 |
| 1002 | 1 | 1 | Α | 3002 |
| 1003 | 1 | 1 | Α | 3003 |
| 1004 | 1 | 1 | В | 3004 |
| 1005 | 1 | 1 | В | 3005 |
| 1006 | 1 | 1 | В | 3006 |
| 1007 | 1 | 1 | С | 3007 |
| 1008 | 1 | 1 | С | 3008 |
| 1009 | 1 | 1 | С | 3009 |

| Statistical Analysis Plan | | | | R-004: Comprehensive <i>in vitro</i> Proarrhythmia Assay<br>) Clinical Phase 1 ECG Biomarker Validation Study |
|---|---|---|---|---|
| 1010 | 1 | 1 | D | 3010 |
| 1011 | 1 | 1 | D | 3011 |
| 1012 | 1 | 1 | D | 3012 |
| 1013 | 1 | 1 | Е | 3013 |
| 1014 | 1 | 1 | Е | 3014 |
| 1015 | 1 | 1 | Е | 3015 |
| 1016 | 1 | 3 | Α | 3016 |
| 1017 | 1 | 3 | Α | 3017 |
| 1018 | 1 | 3 | Α | 3018 |
| 1019 | 1 | 3 | В | 3019 |
| 1020 | 1 | 3 | В | 3020 |
| 1021 | 1 | 3 | В | 3021 |
| 1022 | 1 | 3 | С | 3022 |
| 1023 | 1 | 3 | С | 3023 |
| 1024 | 1 | 3 | С | 3024 |
| 1025 | 1 | 3 | D | 3025 |
| 1026 | 1 | 3 | D | 3026 |
| 1027 | 1 | 3 | D | 3027 |
| 1028 | 1 | 3 | E | 3028 |
| 1029 | 1 | 3 | E | 3029 |
| 1030 | 1 | 3 | E | 3030 |
| 1031 | 1 | 4 | Α | 3031 |
| 1032 | 1 | 4 | Α | 3032 |
| 1033 | 1 | 4 | Α | 3033 |
| 1034 | 1 | 4 | Α | 3034 |
| 1035 | 1 | 4 | В | 3035 |
| 1036 | 1 | 4 | В | 3036 |
| 1037 | 1 | 4 | В | 3037 |
| 1038 | 1 | 4 | В | 3038 |
| 1039 | 1 | 4 | С | 3039 |
| 1040 | 1 | 4 | С | 3040 |
| 1041 | 1 | 4 | С | 3041 |
| 1042 | 1 | 4 | С | 3042 |
| 1043 | 1 | 4 | D | 3043 |

| Statistica | al Analysis | Plan | | R-004: Comprehensive <i>in vitro</i> Proarrhythmia Ass<br>Clinical Phase 1 ECG Biomarker Validation Stu | • |
|---|---|---|---|---|---|
| 1044 | 1 | 4 | D | 3044 | |
| 1045 | 1 | 4 | D | 3045 | |
| 1046 | 1 | 4 | D | 3046 | |
| 1047 | 1 | 4 | E | 3047 | |
| 1048 | 1 | 4 | E | 3048 | |
| 1049 | 1 | 4 | E | 3049 | |
| 1050 | 1 | 4 | E | 3050 | |
| 2001 | 2 | 2 | F-G | 4001 | |
| 2002 | 2 | 2 | F-G | 4002 | |
| 2003 | 2 | 2 | F-G | 4003 | |
| 2004 | 2 | 2 | F-G | 4004 | |
| 2005 | 2 | 2 | F-G | 4005 | |
| 2006 | 2 | 2 | G-F | 4006 | |
| 2007 | 2 | 2 | G-F | 4007 | |
| 2008 | 2 | 2 | G-F | 4008 | |
| 2009 | 2 | 2 | G-F | 4009 | |
| 2010 | 2 | 2 | G-F | 4010 | |

## A.3.1.3 Balanced design summary table

# Print summary table
pander(schedulelong.summary,split.table=Inf)

| PART | SEQ | 1 | 2 | 3 | 4 |
|---|---|---|---|---|---|
| 1 | Α | 1001, 1002,<br>1003 | | 1016, 1017,<br>1018 | 1031, 1032, 1033,<br>1034 |
| 1 | В | 1004, 1005,<br>1006 | | 1019, 1020,<br>1021 | 1035, 1036, 1037,<br>1038 |
| 1 | С | 1007, 1008,<br>1009 | | 1022, 1023,<br>1024 | 1039, 1040, 1041,<br>1042 |
| 1 | D | 1010, 1011,<br>1012 | | 1025, 1026,<br>1027 | 1043, 1044, 1045,<br>1046 |
| 1 | E | 1013, 1014,<br>1015 | | 1028, 1029,<br>1030 | 1047, 1048, 1049,<br>1050 |
| 2 | F-G | | 2001, 2002, 2003, 2004,<br>2005 | | |
| 2 | G-F | | 2006, 2007, 2008, 2009,<br>2010 | | |

#### A.4 Randomization

### A.4.1 Seed random number generator

**TODO:** The unblinded statistician of the sponsor team will be responsible of selecting the seed for the random number generator and update the set.seed statement below accordingly.

```
# Seed the random number generator
myseed <- 123456
set.seed(myseed)
```

#### A.4.2 Randomization schedule code

```
##
# Randomization within blocks by cohort
randomizedschedulelong <- data.frame()</pre>
# Randomize treatment codes within each cohort
for(cohort in unique(schedulelong$COHORT)){
 rsdf <- schedulelong %>% filter(COHORT==cohort)
 # Randomly permute RANDIDs
 rsdf$RANDID <- levels(fct shuffle(as.character(rsdf$RANDID)))</pre>
 rsdf <- rsdf %>% arrange(RANDID)
 randomizedschedulelong <- bind rows(randomizedschedulelong,rsdf)
}
randomizedschedulelong$RANDID <- as.numeric(randomizedschedulelong$RANDID)
randomizedschedulelongwithrplcids <- addpotentialreplacementids(randomizedsch
edulelong)
# Randomization schedule printed in unblinded pharmacist section below
# pander(randomizedschedulelongwithrplcids,split.table=Inf)
```

#### A.4.2.1 Randomized summary table

```
#Format in summary table
randomizedschedulelong.summary <- randomizedschedulelong %>% group_by(COHORT,
SEQ) %>% mutate(RANDIDs=paste0(RANDID,collapse=', ')) %>% select(-RANDID) %>%
ungroup() %>% distinct() %>% spread(COHORT,RANDIDs)
randomizedschedulelong.summary[is.na(randomizedschedulelong.summary)] <- ''
# Randomization summary table printed in unblinded pharmacist section
below
#pander(randomizedschedulelong.summary,split.table=Inf)</pre>
```

#### A.4.2.2 Randomized treatment codes

## A.4.2.3 ## # Randomized treatment codes data.frame ## randomizetreatmentcodes<-F randomizedtreatments <- data.frame()</pre> if (randomizetreatmentcodes){ # Randomize treatment codes within each part for(part in unique(treatments\$PART)){ rtrt <- treatments %>% filter(PART==part) # Randomly permute the levels of the treatment CODEs rtrt\$CODE <- levels(fct\_shuffle(as.character(rtrt\$CODE)))</pre> rtrt <- rtrt %>% arrange(CODE) randomizedtreatments <- bind rows(randomizedtreatments,rtrt)</pre> } } else { randomizedtreatments <- treatments

## A.5 For clinical site unblinded pharmacist

pandoc.header(paste0('The random generator seed was: ', myseed),level=2)

#pander(randomizedtreatments, split.table=Inf)

# Randomized treatment codes printed in unblinded pharmacist

#### A.5.1 The random generator seed was: 123456

#### A.5.2 Randomized treatment codes

TREATMENT

CODE

section below

```
if(randomizetreatmentcodes){
   mystr <- 'Treatments code were randomized\n'
}else{
   mystr <- ('Treatments code as per protocol. Treatment codes NOT randomized\n')
}
sprintf(mystr)
## [1] "Treatments code as per protocol. Treatment codes NOT randomized\n"
pander(randomizedtreatments, split.table=Inf)</pre>
```

PART

```
Α
              Ranolazine
                                  1
  В
              Verapamil
                                  1
  С
          Lopinavir+Ritonavir
                                  1
  D
             Chloroquine
                                  1
  Ε
               Placebo
                                  1
  F
               Dofetilide
                                  2
  G
          Diltiazem+Dofetilide
                                  2
pdf(file = "SCR-004.treatment.codes.pdf")
grid.table(paste0('The random generator seed was: ', myseed, '\n', mystr, '\n
Table in next page'))
grid::grid.newpage()
grid.table(randomizedtreatments, rows=NULL)
dev.off()
## png
##
```

#### A.5.3 Randomization schedule table

pander(randomizedschedulelongwithrplcids,split.table=Inf)

| RANDID | PART | COHORT | SEQ | REPLCMNTID |
|--------|------|--------|-----|------------|
| 1001 | 1 | 1 | С | 3001 |
| 1002 | 1 | 1 | В | 3002 |
| 1003 | 1 | 1 | D | 3003 |
| 1004 | 1 | 1 | В | 3004 |
| 1005 | 1 | 1 | В | 3005 |
| 1006 | 1 | 1 | Α | 3006 |
| 1007 | 1 | 1 | С | 3007 |
| 1008 | 1 | 1 | Ε | 3008 |
| 1009 | 1 | 1 | Ε | 3009 |
| 1010 | 1 | 1 | D | 3010 |
| 1011 | 1 | 1 | Α | 3011 |
| 1012 | 1 | 1 | Α | 3012 |
| 1013 | 1 | 1 | Ε | 3013 |
| 1014 | 1 | 1 | D | 3014 |
| 1015 | 1 | 1 | С | 3015 |
| 1016 | 1 | 3 | С | 3016 |
| 1017 | 1 | 3 | В | 3017 |

| Statistica | ıl Analysis | Plan | | R-004: Comprehensive <i>in vitro</i> Proarrhythmia Assay<br>Clinical Phase 1 ECG Biomarker Validation Study |
|---|---|---|---|---|
| 1018 | 1 | 3 | Α | 3018 |
| 1019 | 1 | 3 | D | 3019 |
| 1020 | 1 | 3 | В | 3020 |
| 1021 | 1 | 3 | E | 3021 |
| 1022 | 1 | 3 | E | 3022 |
| 1023 | 1 | 3 | С | 3023 |
| 1024 | 1 | 3 | В | 3024 |
| 1025 | 1 | 3 | С | 3025 |
| 1026 | 1 | 3 | E | 3026 |
| 1027 | 1 | 3 | D | 3027 |
| 1028 | 1 | 3 | Α | 3028 |
| 1029 | 1 | 3 | Α | 3029 |
| 1030 | 1 | 3 | D | 3030 |
| 1031 | 1 | 4 | E | 3031 |
| 1032 | 1 | 4 | В | 3032 |
| 1033 | 1 | 4 | Α | 3033 |
| 1034 | 1 | 4 | D | 3034 |
| 1035 | 1 | 4 | Α | 3035 |
| 1036 | 1 | 4 | Е | 3036 |
| 1037 | 1 | 4 | С | 3037 |
| 1038 | 1 | 4 | D | 3038 |
| 1039 | 1 | 4 | С | 3039 |
| 1040 | 1 | 4 | D | 3040 |
| 1041 | 1 | 4 | Α | 3041 |
| 1042 | 1 | 4 | В | 3042 |
| 1043 | 1 | 4 | D | 3043 |
| 1044 | 1 | 4 | В | 3044 |
| 1045 | 1 | 4 | E | 3045 |
| 1046 | 1 | 4 | В | 3046 |
| 1047 | 1 | 4 | Α | 3047 |
| 1048 | 1 | 4 | E | 3048 |
| 1049 | 1 | 4 | С | 3049 |
| 1050 | 1 | 4 | C | 3050 |
| 2001 | 2 | 2 | G-F | 4001 |

| Statistical Analysis Plan | SCR-004: Comprehensive in vitro Proarrhythmia Assay |
|---|---|
| | (CiPA) Clinical Phase 1 ECG Biomarker Validation Study |

| 2002 | 2 | 2 | G-F | 4002 |
|------|---|---|-----|------|
| 2003 | 2 | 2 | G-F | 4003 |
| 2004 | 2 | 2 | F-G | 4004 |
| 2005 | 2 | 2 | F-G | 4005 |
| 2006 | 2 | 2 | G-F | 4006 |
| 2007 | 2 | 2 | F-G | 4007 |
| 2008 | 2 | 2 | F-G | 4008 |
| 2009 | 2 | 2 | F-G | 4009 |
| 2010 | 2 | 2 | G-F | 4010 |

```
pdf(file = "SCR-004.randomization.schedule.pdf")
grid.table(paste0('The random generator seed was: ', myseed, '\n Tables by co
hort in next page'))
grid::grid.newpage()
for(cohort in unique(randomizedschedulelongwithrplcids$COHORT)){
    gridExtra::grid.table(randomizedschedulelongwithrplcids %>% filter(COHORT==
    cohort),rows=NULL)
    grid::grid.newpage()
}
dev.off()
## png
## 2
```

#### A.5.4 Randomized summary table

pander(randomizedschedulelong.summary,split.table=Inf)

| PART | SEQ | 1 | 2 | 3 | 4 |
|---|---|---|---|---|---|
| 1 | Α | 1006, 1011,<br>1012 | | 1018, 1028,<br>1029 | 1033, 1035, 1041,<br>1047 |
| 1 | В | 1002, 1004,<br>1005 | | 1017, 1020,<br>1024 | 1032, 1042, 1044,<br>1046 |
| 1 | С | 1001, 1007,<br>1015 | | 1016, 1023,<br>1025 | 1037, 1039, 1049,<br>1050 |
| 1 | D | 1003, 1010,<br>1014 | | 1019, 1027,<br>1030 | 1034, 1038, 1040,<br>1043 |
| 1 | E | 1008, 1009,<br>1013 | | 1021, 1022,<br>1026 | 1031, 1036, 1045,<br>1048 |
| 2 | F-G | | 2004, 2005, 2007, 2008,<br>2009 | | |
| 2 | G-F | | 2001, 2002, 2003, 2006, | | |

2010

## A.6 Appendix: technical information

```
sessionInfo()
## R version 3.3.2 (2016-10-31)
## Platform: x86 64-w64-mingw32/x64 (64-bit)
## Running under: Windows 7 x64 (build 7601) Service Pack 1
##
## locale:
## [1] LC COLLATE=English United States.1252
## [2] LC CTYPE=English United States.1252
## [3] LC MONETARY=English United States.1252
## [4] LC NUMERIC=C
## [5] LC TIME=English United States.1252
##
## attached base packages:
## [1] stats graphics grDevices utils
                                             datasets methods
                                                                bas
е
##
## other attached packages:
## [1] gridExtra 2.2.1 forcats 0.1.1
                                      pander 0.6.0
                                                      dplyr 0.5.0
## [5] purrr_0.2.2 readr_1.0.0
                                      tidyr 0.6.0
                                                      tibble 1.2
## [9] ggplot2_2.2.0 tidyverse_1.0.0
##
## loaded via a namespace (and not attached):
## [1] Rcpp 0.12.7 knitr 1.14
                                        magrittr 1.5
                                                         munsell 0.4
.3
## [5] colorspace 1.2-7 R6 2.2.0
                                        stringr 1.2.0
                                                         plyr 1.8.4
## [9] tools_3.3.2 grid_3.3.2
                                        gtable_0.2.0
                                                         DBI 0.5-1
## [13] htmltools 0.3.5 yaml 2.1.13
                                        lazyeval 0.2.0
                                                         assertthat
0.1
## [17] digest_0.6.12 formatR_1.4
                                        evaluate 0.10
                                                         rmarkdown_1
.1
## [21] stringi_1.1.2 scales_0.4.1
```

## B Step by step example of replacement algorithm

This is just an example of a potential but very unlikely scenario with more than 14 dropouts and with number of dropouts above 20% in at least 2 treatment sequences. In particular, this example shows how replacement will be done with 5 dropouts in the crossover part and 11 dropouts in the parallel part using the randomization schedule example above.

## **B.1** Replacement in crossover part

Potential snapshot of completers and dropouts after Period 1

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Period 1 | Period 2 | Period 3 |
|--------|------|--------|-----|------------|----------|----------|----------|
| 2001 | 2 | 2 | F-G | 4001 | Complete | | |
| 2002 | 2 | 2 | F-G | 4002 | Complete | | |
| 2003 | 2 | 2 | F-G | 4003 | Dropout | | |
| 2004 | 2 | 2 | F-G | 4004 | Dropout | | |
| 2005 | 2 | 2 | F-G | 4005 | Complete | | |
| 2006 | 2 | 2 | G-F | 4006 | Complete | | |
| 2007 | 2 | 2 | G-F | 4007 | Dropout | | |
| 2008 | 2 | 2 | G-F | 4008 | Dropout | | |
| 2009 | 2 | 2 | G-F | 4009 | Dropout | | |
| 2010 | 2 | 2 | G-F | 4010 | Complete | | |

## B.1.1 Move RANDIDs from completers to the next period

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Period 1 | Period 2 | Period 3 |
|---|---|---|---|---|---|---|---|
| 2001 | 2 | 2 | F-G | 4001 | Complete | 2001 | |
| 2002 | 2 | 2 | F-G | 4002 | Complete | 2002 | |
| 2003 | 2 | 2 | F-G | 4003 | Dropout | | |
| 2004 | 2 | 2 | F-G | 4004 | Dropout | | |
| 2005 | 2 | 2 | F-G | 4005 | Complete | 2005 | |
| 2006 | 2 | 2 | G-F | 4006 | Complete | 2006 | |
| 2007 | 2 | 2 | G-F | 4007 | Dropout | | |
| 2008 | 2 | 2 | G-F | 4008 | Dropout | | |
| 2009 | 2 | 2 | G-F | 4009 | Dropout | | |
| 2010 | 2 | 2 | G-F | 4010 | Complete | 2010 | |

## **B.1.2** Replace dropouts

Add one (1) replacement (with lowest RANDID) at a time from each sequence until there are no more replacements to be done or we reach 4 replacements (whichever happens first)

B.1.2.1 Step 1: (replace 2003 from F-G with 4003)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Period 1 | Period 2 | Period 3 |
|--------|------|--------|-----|------------|----------|----------|----------|
| 2001 | 2 | 2 | F-G | 4001 | Complete | 2001 | |
| 2002 | 2 | 2 | F-G | 4002 | Complete | 2002 | |
| 2003 | 2 | 2 | F-G | 4003 | Dropout | 4003 | |
| 2004 | 2 | 2 | F-G | 4004 | Dropout | | |
| 2005 | 2 | 2 | F-G | 4005 | Complete | 2005 | |
| 2006 | 2 | 2 | G-F | 4006 | Complete | 2006 | |
| 2007 | 2 | 2 | G-F | 4007 | Dropout | | |
| 2008 | 2 | 2 | G-F | 4008 | Dropout | | |
| 2009 | 2 | 2 | G-F | 4009 | Dropout | | |
| 2010 | 2 | 2 | G-F | 4010 | Complete | 2010 | |

B.1.2.2 Step 2: (replace 2007 from G-F with 4007)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Period 1 | Period 2 | Period 3 |
|--------|------|--------|-----|------------|----------|----------|----------|
| 2001 | 2 | 2 | F-G | 4001 | Complete | 2001 | |
| 2002 | 2 | 2 | F-G | 4002 | Complete | 2002 | |
| 2003 | 2 | 2 | F-G | 4003 | Dropout | 4003 | |
| 2004 | 2 | 2 | F-G | 4004 | Dropout | | |
| 2005 | 2 | 2 | F-G | 4005 | Complete | 2005 | |
| 2006 | 2 | 2 | G-F | 4006 | Complete | 2006 | |
| 2007 | 2 | 2 | G-F | 4007 | Dropout | 4007 | |
| 2008 | 2 | 2 | G-F | 4008 | Dropout | | |
| 2009 | 2 | 2 | G-F | 4009 | Dropout | | |
| 2010 | 2 | 2 | G-F | 4010 | Complete | 2010 | |

B.1.2.3 Step 3: (replace 2004 from F-G with 4004)

| RA | NDID | PART | COHORT | SEQ | REPLCMNTID | Period 1 | Period 2 | Period 3 |
|---|---|---|---|---|---|---|---|---|
| 2 | 001 | 2 | 2 | F-G | 4001 | Complete | 2001 | |
| 2 | 002 | 2 | 2 | F-G | 4002 | Complete | 2002 | |

| Statistical Analysis Plan | SCR-004: Comprehensive in vitro Proarrhythmia Assay |
|---|---|
| | (CiPA) Clinical Phase 1 ECG Biomarker Validation Study |

| 2003 | 2 | 2 | F-G | 4003 | Dropout | 4003 |
|------|---|---|-----|------|----------|------|
| 2004 | 2 | 2 | F-G | 4004 | Dropout | 4004 |
| 2005 | 2 | 2 | F-G | 4005 | Complete | 2005 |
| 2006 | 2 | 2 | G-F | 4006 | Complete | 2006 |
| 2007 | 2 | 2 | G-F | 4007 | Dropout | 4007 |
| 2008 | 2 | 2 | G-F | 4008 | Dropout | |
| 2009 | 2 | 2 | G-F | 4009 | Dropout | |
| 2010 | 2 | 2 | G-F | 4010 | Complete | 2010 |

## B.1.2.4 Step 4: (replace 2008 from G-F with 4008)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Period 1 | Period 2 | Period 3 |
|--------|------|--------|-----|------------|----------|----------|----------|
| 2001 | 2 | 2 | F-G | 4001 | Complete | 2001 | |
| 2002 | 2 | 2 | F-G | 4002 | Complete | 2002 | |
| 2003 | 2 | 2 | F-G | 4003 | Dropout | 4003 | |
| 2004 | 2 | 2 | F-G | 4004 | Dropout | 4004 | |
| 2005 | 2 | 2 | F-G | 4005 | Complete | 2005 | |
| 2006 | 2 | 2 | G-F | 4006 | Complete | 2006 | |
| 2007 | 2 | 2 | G-F | 4007 | Dropout | 4007 | |
| 2008 | 2 | 2 | G-F | 4008 | Dropout | 4008 | |
| 2009 | 2 | 2 | G-F | 4009 | Dropout | | |
| 2010 | 2 | 2 | G-F | 4010 | Complete | 2010 | |

## **B.1.2.5** End (maximum number of replacements reached)

We have reached the maximum number of replacements (4) for the crossover part, thus we stop adding replacements (subject 2009 is not replaced)

B.2 Replacement in parallel part

Potential snapshot of completers and dropouts after Cohorts 1 and 3 finished.

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status |
|--------|------|--------|-----|------------|----------|
| 1001 | 1 | 1 | Α | 3001 | Complete |
| 1002 | 1 | 1 | Α | 3002 | Dropout |
| 1003 | 1 | 1 | Α | 3003 | Complete |
| 1004 | 1 | 1 | В | 3004 | Dropout |
| 1005 | 1 | 1 | В | 3005 | Complete |
| 1006 | 1 | 1 | В | 3006 | Complete |
| 1007 | 1 | 1 | C | 3007 | Dropout |
| 1008 | 1 | 1 | С | 3008 | Complete |
| 1009 | 1 | 1 | С | 3009 | Complete |
| 1010 | 1 | 1 | D | 3010 | Complete |
| 1011 | 1 | 1 | D | 3011 | Dropout |
| 1012 | 1 | 1 | D | 3012 | Complete |
| 1013 | 1 | 1 | Ε | 3013 | Complete |
| 1014 | 1 | 1 | Ε | 3014 | Dropout |
| 1015 | 1 | 1 | Ε | 3015 | Dropout |
| 1016 | 1 | 3 | Α | 3016 | Complete |
| 1017 | 1 | 3 | Α | 3017 | Complete |
| 1018 | 1 | 3 | Α | 3018 | Dropout |
| 1019 | 1 | 3 | В | 3019 | Dropout |
| 1020 | 1 | 3 | В | 3020 | Complete |
| 1021 | 1 | 3 | В | 3021 | Complete |
| 1022 | 1 | 3 | С | 3022 | Complete |
| 1023 | 1 | 3 | С | 3023 | Complete |
| 1024 | 1 | 3 | С | 3024 | Dropout |
| 1025 | 1 | 3 | D | 3025 | Dropout |
| 1026 | 1 | 3 | D | 3026 | Complete |
| 1027 | 1 | 3 | D | 3027 | Complete |
| 1028 | 1 | 3 | Ε | 3028 | Dropout |
| 1029 | 1 | 3 | Ε | 3029 | Complete |
| 1030 | 1 | 3 | E | 3030 | Complete |

Table of the 10 dropouts to be replaced:

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status |
|--------|------|--------|-----|------------|---------|
| 1002 | 1 | 1 | Α | 3002 | Dropout |
| 1004 | 1 | 1 | В | 3004 | Dropout |
| 1007 | 1 | 1 | С | 3007 | Dropout |
| 1011 | 1 | 1 | D | 3011 | Dropout |
| 1014 | 1 | 1 | Ε | 3014 | Dropout |
| 1015 | 1 | 1 | Ε | 3015 | Dropout |
| 1018 | 1 | 3 | Α | 3018 | Dropout |
| 1019 | 1 | 3 | В | 3019 | Dropout |
| 1024 | 1 | 3 | С | 3024 | Dropout |
| 1025 | 1 | 3 | D | 3025 | Dropout |
| 1028 | 1 | 3 | Ε | 3028 | Dropout |

## **B.2.1 Step 1: (replace subject 1014 from placebo)**

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | |
| 1004 | 1 | 1 | В | 3004 | Dropout | |
| 1007 | 1 | 1 | С | 3007 | Dropout | |
| 1011 | 1 | 1 | D | 3011 | Dropout | |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Ε | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | |
| 1019 | 1 | 3 | В | 3019 | Dropout | |
| 1024 | 1 | 3 | С | 3024 | Dropout | |
| 1025 | 1 | 3 | D | 3025 | Dropout | |
| 1028 | 1 | 3 | Ε | 3028 | Dropout | |

**B.2.2** Step 2: (replace subject 1002 from ranolazine)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | |
| 1007 | 1 | 1 | С | 3007 | Dropout | |
| 1011 | 1 | 1 | D | 3011 | Dropout | |

| Statistical Analysis Plan | SCR-004: Comprehensive in vitro Proarrhythmia Assay |
|---|---|
| | (CiPA) Clinical Phase 1 ECG Biomarker Validation Study |

| 3014 | Dropout | 3014 | Е | 1 | 1 | 1014 |
|------|---------|------|---|---|---|------|
| | Dropout | 3015 | E | 1 | 1 | 1015 |
| | Dropout | 3018 | Α | 3 | 1 | 1018 |
| | Dropout | 3019 | В | 3 | 1 | 1019 |
| | Dropout | 3024 | С | 3 | 1 | 1024 |
| | Dropout | 3025 | D | 3 | 1 | 1025 |
| | Dropout | 3028 | E | 3 | 1 | 1028 |

# **B.2.3** Step 3: (replace subject 1004 from verapamil)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | С | 3007 | Dropout | |
| 1011 | 1 | 1 | D | 3011 | Dropout | |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Ε | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | |
| 1019 | 1 | 3 | В | 3019 | Dropout | |
| 1024 | 1 | 3 | С | 3024 | Dropout | |
| 1025 | 1 | 3 | D | 3025 | Dropout | |
| 1028 | 1 | 3 | Ε | 3028 | Dropout | |

## **B.2.4** Step 4: (replace subject 1011 from chloroquine)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | С | 3007 | Dropout | |
| 1011 | 1 | 1 | D | 3011 | Dropout | 3011 |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Ε | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | |
| 1019 | 1 | 3 | В | 3019 | Dropout | |
| 1024 | 1 | 3 | С | 3024 | Dropout | |

| Statistical Analysis Plan | SCR-004: Comprehensive in vitro Proarrhythmia Assay |
|---|---|
| | (CiPA) Clinical Phase 1 ECG Biomarker Validation Study |

| 1025 | 1 | 3 | D | 3025 | Dropout |
|------|---|---|---|------|---------|
| 1028 | 1 | 3 | Ε | 3028 | Dropout |

## **B.2.5** Step 5: (replace subject 1007 from lopinavir+ritonavir)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | С | 3007 | Dropout | 3007 |
| 1011 | 1 | 1 | D | 3011 | Dropout | 3011 |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Ε | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | |
| 1019 | 1 | 3 | В | 3019 | Dropout | |
| 1024 | 1 | 3 | С | 3024 | Dropout | |
| 1025 | 1 | 3 | D | 3025 | Dropout | |
| 1028 | 1 | 3 | Ε | 3028 | Dropout | |

## B.2.6 Step 6: (replace subject 1028 from placebo)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | С | 3007 | Dropout | 3007 |
| 1011 | 1 | 1 | D | 3011 | Dropout | 3011 |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Ε | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | |
| 1019 | 1 | 3 | В | 3019 | Dropout | |
| 1024 | 1 | 3 | С | 3024 | Dropout | |
| 1025 | 1 | 3 | D | 3025 | Dropout | |
| 1028 | 1 | 3 | Ε | 3028 | Dropout | 3028 |

## **B.2.7 Step 7: (replace subject 1018 from ranolazine)**

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|--------|-------------|
|--------|------|--------|-----|------------|--------|-------------|

| Statistical Analysis Plan | SCR-004: Comprehensive in vitro Proarrhythmia Assay |
|---|---|
| | (CiPA) Clinical Phase 1 ECG Biomarker Validation Study |

| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
|------|---|---|---|------|---------|------|
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | С | 3007 | Dropout | 3007 |
| 1011 | 1 | 1 | D | 3011 | Dropout | 3011 |
| 1014 | 1 | 1 | E | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Е | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | 3018 |
| 1019 | 1 | 3 | В | 3019 | Dropout | |
| 1024 | 1 | 3 | С | 3024 | Dropout | |
| 1025 | 1 | 3 | D | 3025 | Dropout | |
| 1028 | 1 | 3 | Е | 3028 | Dropout | 3028 |

# B.2.8 Step 8: (replace subject 1019 from verapamil)

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | C | 3007 | Dropout | 3007 |
| 1011 | 1 | 1 | D | 3011 | Dropout | 3011 |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Ε | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | 3018 |
| 1019 | 1 | 3 | В | 3019 | Dropout | 3019 |
| 1024 | 1 | 3 | С | 3024 | Dropout | |
| 1025 | 1 | 3 | D | 3025 | Dropout | |
| 1028 | 1 | 3 | Ε | 3028 | Dropout | 3028 |

## **B.2.9 Step 9: (replace subject 1025 from chloroquine)**

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | С | 3007 | Dropout | 3007 |
| 1011 | 1 | 1 | D | 3011 | Dropout | 3011 |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |

| Statistical Analysis Plan | | | | SCR-004: Comprehensive <i>in vitro</i> Proarrhythmia Assay (CiPA) Clinical Phase 1 ECG Biomarker Validation Study | | |
|---|---|---|---|---|---|---|
| 1015 | 1 | 1 | E | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | 3018 |
| 1019 | 1 | 3 | В | 3019 | Dropout | 3019 |

3024

3025

3028

Dropout

Dropout

Dropout

3025

3028

B.2.10 Step 10: (replace subject 1024 from lopinavir+ritonavir)

С

D

Ε

1024

1025

1028

1

1

1

3

3

3

| RANDID | PART | COHORT | SEQ | REPLCMNTID | Status | Replacement |
|--------|------|--------|-----|------------|---------|-------------|
| 1002 | 1 | 1 | Α | 3002 | Dropout | 3002 |
| 1004 | 1 | 1 | В | 3004 | Dropout | 3004 |
| 1007 | 1 | 1 | С | 3007 | Dropout | 3007 |
| 1011 | 1 | 1 | D | 3011 | Dropout | 3011 |
| 1014 | 1 | 1 | Ε | 3014 | Dropout | 3014 |
| 1015 | 1 | 1 | Ε | 3015 | Dropout | |
| 1018 | 1 | 3 | Α | 3018 | Dropout | 3018 |
| 1019 | 1 | 3 | В | 3019 | Dropout | 3019 |
| 1024 | 1 | 3 | С | 3024 | Dropout | 3024 |
| 1025 | 1 | 3 | D | 3025 | Dropout | 3025 |
| 1028 | 1 | 3 | Ε | 3028 | Dropout | 3028 |

## B.2.11 Step 11: End (maximum number of 14 replacements reached)

We have reached the maximum number of replacements (14) for the study, thus we stop adding replacements (subject 1015 is not replaced in this example)